CLINICAL TRIAL: NCT02402894
Title: Follow-up of Person-centered Care of Young Adults With Rheumatic Disease Uppföljning av Personcentrerat omhändertagande av Unga Vuxna Med Reumatisk Sjukdom (Unga-vuxna Studien) (Swedish)
Brief Title: Follow-up of Person-centered Care of Young Adults With Rheumatic Disease
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014-10-08
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2022-04

CONDITIONS: Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
The purpose of the study is to study how a person-centered structured team caretaking of young adults (16-23 years) with newly diagnosed rheumatoid arthritis (RA), spondartrit (SpA) and psoriasartrit (PsA) in routine clinical care affect and predict the patient's health and ability to manage their everyday lives. Also included in the project is a long-term follow-up (up to 50 years) where the investigators want to investigate factors predicting good general health, low disease activity, good physical function, and comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* 16-23 years
* newly diagnosed RA according to the ACR / EULAR 2010 criteria, SpA according to CASPAR criteria, or AS according to the ASAS criteria.
* Ability to understand the Swedish language in speech and writing.

Exclusion Criteria:

* Existing rheumatic disease
* Other healthcare demanding serious illness

Ages: 16 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young adults (16-23 years) with newly diagnosed rheumatoid arthritis (RA), spondartrit (SpA) and psoriasartrit (PsA) in routine clinical care. In total 100 patients, no healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
General health as measured by VAS | This study consists of a 1-year primary study and a long term follow-up (up to 50 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Reumatology, Sahlgrenska University Hospital, VastraGotaland, Gothenburg, Sweden